CLINICAL TRIAL: NCT01058460
Title: A Randomized Controlled Trial Comparing Concomitant HPV-cytology Testing With Conventional Cytology Testing for the Detection of High Grade Cervical Intraepithelial Neoplasia in Primary Cervical Cancer Screening in Hong Kong
Brief Title: HPV-cytology Testing Versus Cytology Testing for the Detection of High Grade CIN
Acronym: COCY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Family Planning Association of Hong Kong (Other)
Responsible Party: Professor Hextan Y.S. Ngan, Department of Obstetrics & Gynaecology, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UW09-377
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia
Keywords: Cervical Intraepithelial Neoplasia, Grade III; Cervical Intraepithelial Neoplasia, Grade II
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- cytology (No Intervention): Subjects in the control arm will receive conventional cytology testing and HPV testing at baseline. Follow up management will be based on the cytology result according to current practice.
- HPV-cytology (Experimental): Subjects in the HPV-cytology arm will receive HPV testing and cytology testing at baseline. Follow up management will be based on both results.
  Interventions: Procedure: HPV-cytology co-testing

INTERVENTIONS:
Procedure: HPV-cytology co-testing — Subjects will receive HPV testing and conventional cytology testing at baseline. Follow up management will be based on both results.
  Arms: HPV-cytology

SUMMARY:
To compare the effects of conventional cytology testing with concommitant HPV-cytology testing for the detection of high grade cervical lesions in primary cervical cancer screening in Hong Kong

Hypotheses:

1. There is a significant difference in the number of CIN2+ cases detected between the cytology testing group and the cytology-HPV co-testing group at baseline.
2. Significantly more CIN2+ cases will be detected at the second round of screening among participants with normal cytology result in the control arm than those with normal cytology and negative HPV results in the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese women aged 30 to 60 years who have completed a written consent
* Women who have not attended screening for the past 3 years or more will be given priority

Exclusion Criteria:

* Currently pregnant
* Without a cervix
* Congenital abnormalities of the lower genital tract
* Previous history of invasive cervical cancer
* Who has been followed-up or treated for an abnormal cytology result in the past 12 months
* Who are unable to provide consent

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12000 (Estimated)
Dates: Start 2010-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Histological CIN2, CIN3 and cervical carcinoma | At baseline and each subsequent follow-up

SECONDARY OUTCOMES:
Clearance of mild cervical abnormalities among HPV negative subjects | At baseline and 1-year after

CONTACTS AND LOCATIONS:
Overall Officials: Hextan YS Ngan, MD, MBBS, Principal Investigator — Department of Obstetrics & Gynaecology, The University of Hong Kong
Locations (1):
- Department of Obstetrics & Gynaecology, The University of Hong Kong, Hong Kong SAR, China